CLINICAL TRIAL: NCT03702998
Title: Incidence and Mortality of Hepatocellular Carcinoma in HIV-infected Individuals in an Asian Population
Brief Title: Hepatocellular Carcinoma in HIV-infected Individuals in Asian Population
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: HCC_HIV protocol_V3_26042017
Record Dates: First submitted 2018-07-09; First posted 2018-10-11 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections; Hepatitis B; Hepatitis C; Hepatocellular Carcinoma
MeSH Terms: conditions — HIV Infections; Hepatitis B; Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV-infected individuals +/- HBV/ HCV: 1 All HIV-infected individuals followed up in all public HIV clinics with and without HBV and/or HCV co-infection will be included in the analysis.
  1.1 Inclusion criteria for HIV-infected individuals with and without HBV or HCV co-infection: 1.1.1 Positive HIV antibody 1.1.2 At least one visit in one of the HIV clinics 1.1.3 Subjects with positive HBsAg and/or anti-HBc will be regarded as having HBV co-infection 1.1.4 Subjects with positive HCV antibody will be regarded as having HCV co-infection
- HBV/HCV mono-infected individuals: 2 All HBV and/or HCV-infected individuals followed up in public hospitals will be identified from the Hospital Authority electronic database.
  2.1 Inclusion criteria for HBV/HCV mono-infected individuals 2.1.1 Documented diagnosis of hepatitis B or hepatitis C infection, or 2.1.2 Positive HBsAg and/or anti-HBc, or 2.1.3 Positive HCV antibody, and 2.1.4 Negative HIV antibody result, or no record of HIV diagnosis or anti-retroviral therapy prescription

SUMMARY:
This is a retrospective study, all HIV-infected individuals followed up at the three designated HIV clinics in Hong Kong with and without HBV and/or HCV co-infection will be included in the analysis. The incidence and mortality of HCC among HIV-infected individuals with and without HBV/HCV co-infection in an Asian population will be determined.

DETAILED DESCRIPTION:
The incidence of hepatocellular carcinoma (HCC) is increasing over time among the HIV-infected population, and is an increasingly important cause of morbidity and mortality in HIV-infected individuals. Despite effective treatment for HBV and HCV infections, HCC is still reported in treated HIV-infected individuals with HBV/HCV co-infections. Currently, data on the risk and outcomes of HCC in HIV infected populations in Asia is lacking. This study aims to evaluate the incidence of HCC in HIV-infected individuals with and without HBV/HCV co-infection, and HBV/HCV mono-infected individuals in Hong Kong.

This is a retrospective study, all HIV-infected individuals followed up at the three designated HIV clinics in Hong Kong with and without HBV and/or HCV co-infection will be included in the analysis. The burden of HCC among HIV-infected individuals with and without HBV/HCV co-infection in an Asian population will be determined by comparing their incidence and mortality.

Objectives:

1. To determine the burden of HCC among HIV-infected individuals with and without HBV/HCV co-infection in an Asian population
2. To compare the incidence of HCC between HIV-infected individuals with HBV/HCV co-infection and HIV-uninfected individuals with HBV or HCV-monoinfection
3. To compare the mortality rate of HCC between HIV-infected individuals with HBV/HCV co- infection and HIV-uninfected individuals with HBV or HCV-monoinfection.

Study procedures

1. The electronic databases and medical records of all three HIV centres, and Clinical Data Analysis and Reporting System (CDARS) will be reviewed for data extraction for HIV-infected individuals.
2. The medical records and electronic database of Hospital Authority, Clinical Data Analysis and Reporting System (CDARS), will be reviewed for data extraction for HBV and HCV-infected individuals without HIV infection.
3. The following demographic and clinical data will be retrieved:

3.1 Date of birth, gender, ethnicity 3.2 Date of diagnosis of HIV infection 3.3 Route of transmission of HIV infection 3.4 Other concomitant chronic liver diseases (including alcoholic liver disease, fatty liver, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis etc) 3.5 Presence of cirrhosis and cirrhotic complications (including ascites, esophageal varices, encephalopathy, hepatorenal syndrome, hepatic coma) 3.6 Other comorbidities, including diabetes mellitus, drug-induced hepatitis, alcoholism 3.7 History of AIDS-defining illness 3.8 Nadir CD4 count, latest CD4 count 3.9 Latest HIV viral load 3.10 Bilirubin, ALT, ALP, total protein, albumin, platelet count, prothrombin time 3.11 HBeAg, anti-HBe, HBV DNA, HCV RNA 3.12 Antiviral therapy for HIV, HBV and HCV, including date of initiation and cessation, and name of drugs prescribed 3.13 Date of last follow-up 3.14 Date of diagnosis of liver cancer 3.15 Treatment of liver cancer (surgical, locoregional, chemotherapy, others) 3.16 Date and cause of death

ELIGIBILITY:
1. HIV-infected individuals with and without HBV or HCV co-infection:

   Inclusion criteria:
   * Positive HIV antibody
   * At least one visit in one of the HIV clinics
   * Subjects with positive HBsAg and/or anti-HBc will be regarded as having HBV co-infection
   * Subjects with positive HCV antibody will be regarded as having HCV co-infection

   Exclusion criteria:

   -nil
2. HBV/HCV mono-infected individuals:

Inclusion criteria:

* Documented diagnosis of hepatitis B or hepatitis C infection, or
* Positive HBsAg and/or anti-HBc, or
* Positive HCV antibody, and
* Negative HIV antibody result, or no record of HIV diagnosis or anti-retroviral therapy prescription

Exclusion criteria:

- nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected individuals with and without HBV/HCV co-infection, and HBV/HCV mono-infected individuals in Hong Kong
Sampling Method: Probability Sample
Enrollment: 3900 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Incidence of HCC | From the time of diagnosis up to 20 years of follow up.
  Diagnoses that will be included in the primary outcome include: ICD9 coded diagnoses of cancer of liver (155); malignant neoplasm of liver, primary (155.0); cancer of liver, primary (155.0(0)), primary carcinoma of liver (155.0(1)); hepatocellular carcinoma (155.0(2)); malignant neoplasm of liver, not specified (155.2); cancer of liver (155.2(0)); carcinoma of liver (155.2(1)).

SECONDARY OUTCOMES:
Mortality due to HCC or liver-related conditions | From the time of diagnosis up to 20 years of follow up.
  1. Cause of death as documented in death certificate that included HCC as primary or secondary causes of death will be regarded as death due to HCC.
  2. Cause of death due to liver-related conditions will include the following conditions: hepatitis B, hepatitis C, viral hepatitis, hepatic failure, chronic hepatitis, cirrhosis of liver, liver failure, chronic liver disease, or hepatorenal syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lui, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong